CLINICAL TRIAL: NCT01106794
Title: Molecular Analysis of Samples From Patients With Diffuse Intrinsic Pontine Glioma and Brainstem Glioma
Status: Recruiting | Type: Observational
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Javad Nazarian, Associate Professor, Children's National Research Institute
Other Study IDs: DIPG-1
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Brainstem Glioma
Keywords: diffuse intrinsic pontine glioma; DIPG; childhood brainstem glioma; pediatric brainstem glioma; brainstem glioma; BSG
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid, serum, urine, brainstem tumor and constitutional tissue from patients with diffuse intrinsic pontine glioma or brainstem glioma will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient samples: Fresh-frozen and fixed tumor samples, correspondent normal brain tissue samples, cerebrospinal fluid, urine, and serum samples from patients affected with diffuse intrinsic pontine glioma or brainstem glioma

SUMMARY:
The purpose of this study is to prospectively collect specimens from pediatric patients with diffuse intrinsic pontine glioma or brainstem glioma, either during therapy or at autopsy, in order to characterize the molecular abnormalities of this tumor.

DETAILED DESCRIPTION:
High grade diffuse intrinsic pontine glioma (DIPG) accounts for approximately 80% of pediatric brainstem tumors and 10% of pediatric brain tumors, and is the most lethal form of brainstem gliomas in children. There is currently no effective therapy to treat these tumors. We hypothesize that this tumor exhibits unique molecular abnormalities leading to altered RNA and protein expression. The aim of this trial is to collect specimens from pediatric patients with diffuse intrinsic pontine glioma including serum, cerebrospinal fluid, urine, brain tumor and other constitutional tissue, during therapy and/or at autopsy. Our goal is to study this tissue to characterize the genetic abnormalities that lead to tumor formation in order to identify key molecules as biomarkers which we can target to design and test new and more effective treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age with clinical and radiologic diagnosis of diffuse intrinsic pontine glioma
* Patients with other high-grade gliomas originating in the brainstem
* Patients with focal gliomas (WHO grade I/II) of the brainstem

Exclusion Criteria:

* Patients with any type of infiltrative low grade (WHO grade I and II) or high grade glioma (WHO grade III and IV) originating outside the brainstem
* Patients harboring primary brainstem tumors with other histologic diagnoses (e.g., PNET)

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-04 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Genome-wide expression patterns of RNA in tumor samples, normal brainstem tissue and cerebrospinal fluid using Affymetrix gene expression profiling | 5 years
  Collected tumor and normal samples will potentially be used for RNA genome-wide expression pattern profiling.
Validation of results of the genome-wide analysis | 5 years
  The molecular analysis done on collected samples will be validated through whole genome sequencing.
Proteomic profiling of tumor, normal brainstem tissue and cerebrospinal fluid | 5 years
  To obtain full characterization of collected samples, proteomic profiling will be done on tumor and normal samples collected.
Protein expression patterns as assessed by immunohistochemistry and western blot compared to normal brainstem tissue | 5 years
  Collected tumor and normal samples will have the immunochemistry and western blot compared to assess protein expression variation.
Genome-wide analysis of tumor samples and normal brainstem tissue | 5 years
  To obtain full characterization of collected samples, whole genome sequencing will be done on tumor and normal samples collected.
In vitro and in vivo molecular analysis of collected samples | 5 years
  Collected samples will potentially be used for in vitro analysis and generation of animal models of this tumor.

SECONDARY OUTCOMES:
Assess aspects associated with specimen acquisition, including potential benefits and drawbacks | 5 years
  In an effort to continue to draw knowledge from samples collected, potential benefits and drawbacks from specimen acquisition will be continuously accessed.

CONTACTS AND LOCATIONS:
Overall Officials: Javad Nazarian, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Becher OJ, Hambardzumyan D, Walker TR, Helmy K, Nazarian J, Albrecht S, Hiner RL, Gall S, Huse JT, Jabado N, MacDonald TJ, Holland EC. Preclinical evaluation of radiation and perifosine in a genetically and histologically accurate model of brainstem glioma. Cancer Res. 2010 Mar 15;70(6):2548-57. doi: 10.1158/0008-5472.CAN-09-2503. Epub 2010 Mar 2. PMID 20197468
- [Background] Panditharatna E, Yaeger K, Kilburn LB, Packer RJ, Nazarian J. Clinicopathology of diffuse intrinsic pontine glioma and its redefined genomic and epigenomic landscape. Cancer Genet. 2015 Jul-Aug;208(7-8):367-73. doi: 10.1016/j.cancergen.2015.04.008. Epub 2015 May 1. PMID 26206682
- [Background] Yadavilli S, Scafidi J, Becher OJ, Saratsis AM, Hiner RL, Kambhampati M, Mariarita S, MacDonald TJ, Codispoti KE, Magge SN, Jaiswal JK, Packer RJ, Nazarian J. The emerging role of NG2 in pediatric diffuse intrinsic pontine glioma. Oncotarget. 2015 May 20;6(14):12141-55. doi: 10.18632/oncotarget.3716. PMID 25987129
- [Background] Kambhampati M, Perez JP, Yadavilli S, Saratsis AM, Hill AD, Ho CY, Panditharatna E, Markel M, Packer RJ, Nazarian J. A standardized autopsy procurement allows for the comprehensive study of DIPG biology. Oncotarget. 2015 May 20;6(14):12740-7. doi: 10.18632/oncotarget.3374. PMID 25749048
- [Background] Kambhampati M, Panditharatna E, Yadavilli S, Saoud K, Lee S, Eze A, Almira-Suarez MI, Hancock L, Bonner ER, Gittens J, Stampar M, Gaonkar K, Resnick AC, Kline C, Ho CY, Waanders AJ, Georgescu MM, Rance NE, Kim Y, Johnson C, Rood BR, Kilburn LB, Hwang EI, Mueller S, Packer RJ, Bornhorst M, Nazarian J. Harmonization of postmortem donations for pediatric brain tumors and molecular characterization of diffuse midline gliomas. Sci Rep. 2020 Jul 2;10(1):10954. doi: 10.1038/s41598-020-67764-2. PMID 32616776
- [Result] Ballester LY, Wang Z, Shandilya S, Miettinen M, Burger PC, Eberhart CG, Rodriguez FJ, Raabe E, Nazarian J, Warren K, Quezado MM. Morphologic characteristics and immunohistochemical profile of diffuse intrinsic pontine gliomas. Am J Surg Pathol. 2013 Sep;37(9):1357-64. doi: 10.1097/PAS.0b013e318294e817. PMID 24076776
- [Result] Saratsis AM, Yadavilli S, Magge S, Rood BR, Perez J, Hill DA, Hwang E, Kilburn L, Packer RJ, Nazarian J. Insights into pediatric diffuse intrinsic pontine glioma through proteomic analysis of cerebrospinal fluid. Neuro Oncol. 2012 May;14(5):547-60. doi: 10.1093/neuonc/nos067. Epub 2012 Apr 5. PMID 22492959
- [Result] Ahsan S, Raabe EH, Haffner MC, Vaghasia A, Warren KE, Quezado M, Ballester LY, Nazarian J, Eberhart CG, Rodriguez FJ. Increased 5-hydroxymethylcytosine and decreased 5-methylcytosine are indicators of global epigenetic dysregulation in diffuse intrinsic pontine glioma. Acta Neuropathol Commun. 2014 Jun 3;2:59. doi: 10.1186/2051-5960-2-59. PMID 24894482
- [Result] Buczkowicz P, Hoeman C, Rakopoulos P, Pajovic S, Letourneau L, Dzamba M, Morrison A, Lewis P, Bouffet E, Bartels U, Zuccaro J, Agnihotri S, Ryall S, Barszczyk M, Chornenkyy Y, Bourgey M, Bourque G, Montpetit A, Cordero F, Castelo-Branco P, Mangerel J, Tabori U, Ho KC, Huang A, Taylor KR, Mackay A, Bendel AE, Nazarian J, Fangusaro JR, Karajannis MA, Zagzag D, Foreman NK, Donson A, Hegert JV, Smith A, Chan J, Lafay-Cousin L, Dunn S, Hukin J, Dunham C, Scheinemann K, Michaud J, Zelcer S, Ramsay D, Cain J, Brennan C, Souweidane MM, Jones C, Allis CD, Brudno M, Becher O, Hawkins C. Genomic analysis of diffuse intrinsic pontine gliomas identifies three molecular subgroups and recurrent activating ACVR1 mutations. Nat Genet. 2014 May;46(5):451-6. doi: 10.1038/ng.2936. Epub 2014 Apr 6. PMID 24705254
- [Result] Saratsis AM, Kambhampati M, Snyder K, Yadavilli S, Devaney JM, Harmon B, Hall J, Raabe EH, An P, Weingart M, Rood BR, Magge SN, MacDonald TJ, Packer RJ, Nazarian J. Comparative multidimensional molecular analyses of pediatric diffuse intrinsic pontine glioma reveals distinct molecular subtypes. Acta Neuropathol. 2014;127(6):881-95. doi: 10.1007/s00401-013-1218-2. Epub 2013 Dec 3. PMID 24297113
- [Result] Nikbakht H, Panditharatna E, Mikael LG, Li R, Gayden T, Osmond M, Ho CY, Kambhampati M, Hwang EI, Faury D, Siu A, Papillon-Cavanagh S, Bechet D, Ligon KL, Ellezam B, Ingram WJ, Stinson C, Moore AS, Warren KE, Karamchandani J, Packer RJ, Jabado N, Majewski J, Nazarian J. Spatial and temporal homogeneity of driver mutations in diffuse intrinsic pontine glioma. Nat Commun. 2016 Apr 6;7:11185. doi: 10.1038/ncomms11185. PMID 27048880
- See also: Children's National Medical Center — https://childrensnational.org/research